CLINICAL TRIAL: NCT00212758
Title: IGF-1 Generation Test in Children With Chronic Kidney Disease
Brief Title: A Study to Optimize Growth Hormone Dosing in Children With Chronic Kidney Disease by Measuring IGF-1 Levels in Blood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Amira Al-Uzri, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Genentech # 303-MO1
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Kidney Failure, Chronic; Growth Hormone Deficiency
Keywords: Short stature; children; kidney failure, chronic; Growth
MeSH Terms: conditions — Kidney Failure, Chronic; Dwarfism, Pituitary; Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low- Standard GH dose (Active Comparator): This arm will receive Low dose of growth hormone (GH) (Nutropin AQ), for 7 days in a cross over design. Low dose GH will be 0.025 mg/kg/day. This will be followed by 2 weeks of wash out, then subjects will receive and the standard dose of Nutropin AQ (GH) at 0.05 mg/kg/dose given subcutaneously for another 7 days. IGF-I levels are measured after 7 days of the Low and the Standard dose of GH. After that all subjects will be treated with the standard dose of GH therapy of 0.05 mg/kg/day for 6 months and re-evaluated. If growth is adequate then subjects will continue on standard dose of GH for another 6 months for a total of 12 months.
  Interventions: Drug: Nutropin AQ
- Standard-Low GH dose (7 Days) (Active Comparator): This arm will receive Standard dose of growth hormone (GH) (Nutropin AQ), for 7 days in a cross over design. Standard dose GH will be 0.5 mg/kg/day. This will be followed by 2 weeks of wash out, then subjects will receive and the Low dose of Nutropin AQ (GH) at 0.025 mg/kg/dose given subcutaneously for another 7 days. IGF-I levels are measured after 7 days of the Low and the Standard dose of GH. After that all subjects will be treated with the standard dose of GH therapy of 0.05 mg/kg/day for 6 months and re-evaluated. If growth is adequate then subjects will continue on standard dose of GH for another 6 months for a total of 12 months.
  Interventions: Drug: Nutropin AQ

INTERVENTIONS:
Drug: Nutropin AQ — Nutropin AQ
  Other Names: Growth hormone

SUMMARY:
Treatment with growth hormone (GH; a hormone made by the body that stimulates growth) has been shown to be helpful in treating children with chronic kidney disease who fail to grow. The amount of growth that is seen in children treated with growth hormone varies widely for unknown reasons. Growth hormone works by producing another hormone in the liver called insulin-like growth factor-1, or IGF-1 for short. IGF-1 stimulates the bones to grow. The amount of IGF-1 in the blood may directly affect the amount of growth in each child. At this time, growth hormone therapy in children depends on giving a certain dose of growth hormone for each child based on his or her weight. If after 3-6 months on this dose of growth hormone the change in height is not enough, then the dose of growth hormone is increased until enough growth is seen. This method of dosing of growth hormone may take a long time and is complicated and time-consuming.

The purpose of this study is to measure the amount of IGF-1 produced by the body as a result of giving 2 different doses of growth hormone in children for 7 days only. The study investigator hopes to find the most favorable level of IGF-1 generated after 7 days of growth hormone that correlates with good growth of children with kidney disease. Then instead of dosing growth hormone by weight, like is done now, researchers can dose growth hormone by the amount of IGF-1 that the body produces. Being able to dose more effectively will save valuable time for the child to grow and will shorten the overall duration of growth hormone therapy.

The investigators will also determine the effect of inflammatory cytokines Il-6 and TNF-alpha on growth hormone insensitivity and hence IGF-1 generation test in the same population.

DETAILED DESCRIPTION:
The study will involve 30 children with chronic kidney disease and failure to grow. The study will last for 14 months. There will be a screening clinic visit if the child qualifies for the study, Week -8. Each clinic visit will include, getting a medical history, a physical exam, and a blood test. Also an x-ray of the wrist to calculate bone age. If abnormal blood values are found as a result of kidney failure then an attempt will be made to correct them over the next 2 months before enrollment in the study.

Also children will be asked to keep track of all of the foods for 3 days every month during the study. A study nutritionist will call them once each month to go over the food diary.

At study Week -4, children will come again for a clinic visit. Then at Week 0 of the study, a decision will be made randomly based on the level of kidney function to what dose of growth hormone a child will receive. This will be either a low dose of growth hormone or a high dose of growth hormone.

At the Week 1 and Week 4 visits, children will come for a clinic visit. Children will take growth hormone (through a needle under the skin) every night for a full 7 days during each of the two weeks. In the mornings before the 1st and after the 7th dose both weeks, children will have their blood drawn to check IGF-1 levels.

During Weeks 2 and 3, children will not take any growth hormone in order to allow the body to clear, or "wash-out", the medication from the system before Week 4.

At Week 5, children will begin taking growth hormone each evening and continue to do so every day through Week 28. Then, for Weeks 29 and 30, children will have another "wash-out" period with no growth hormone treatment.

At Week 31, blood will be drawn in the mornings before the 1st and after the 7th dose of growth hormone treatment. From Week 32 on, children will take growth hormone every evening and continue to do so through Week 56, the end of the study.

Also at week 1, skin fold measurements to assess body fat will be done on all subjects. A DEXA scan, a test that measures body fat and muscle mass will be done on the older children in the study on an optional basis on Weeks 1, 28 and 56. Another wrist X-ray for bone age will be repeated at 56 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 2-18 years of age with chronic renal failure.
* Estimated creatinine clearance between 25-75 ml/min/1.73 m2 calculated by the Schwartz formula.
* Height standard deviation score (SDS) more than -1.88 or annual height velocity SD of more than -2.0 for age and sex for the preceding 6 months.
* No history of growth hormone therapy.
* Cystinosis subjects may qualify for the study if they meet other inclusion criteria and have an estimated creatinine clearance of 25-75 ml/min/1.73 m2.
* Bone age less than 16 years for boys and less than 13 years for girls.
* Subjects with chronic kidney failure who are off steroid therapy or other drugs that interfere with growth for at least 6 months.

Exclusion Criteria:

* Subjects on dialysis and kidney transplant recipients.
* Patients with significant renal osteodystrophy or an intact parathyroid (PTH) level more than 500 pg/ml over the last 3 months prior to enrollment.
* Diabetes mellitus.
* History of malignancy.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amira Y Al-Uzri, M.D., Principal Investigator — Oregon Health and Science University
Locations (8):
- United States (8):
  - Loma Linda UMC & Children's Hospital, Loma Linda, California
  - University of California in Los Angeles (UCLA), Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Texas Children's Hospital, Houston, Texas
  - UT Houston Medical School, Houston, Texas
  - University of Washington, Children's Hospital & Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Buckway CK, Guevara-Aguirre J, Pratt KL, Burren CP, Rosenfeld RG. The IGF-I generation test revisited: a marker of GH sensitivity. J Clin Endocrinol Metab. 2001 Nov;86(11):5176-83. doi: 10.1210/jcem.86.11.8019. PMID 11701674
- [Derived] Al-Uzri A, Swinford RD, Nguyen T, Jenkins R, Gunsul A, Kachan-Liu SS, Rosenfeld R. The utility of the IGF-I generation test in children with chronic kidney disease. Pediatr Nephrol. 2013 Dec;28(12):2323-33. doi: 10.1007/s00467-013-2570-0. Epub 2013 Sep 7. PMID 24013497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter trial. Patients were recruited from pediatric nephrology clinics at various centers.
Pre-assignment Details: A two month run-in period was implemented to stabilize subjects and correct any metabolic abnormalities that may affect growth. This two month period may be waived per the center PI if patient was deemed stable. Patients were randomized to either a low or standard dose of GH (Nutropin AQ)used in the IGF-I generation.
Groups:
- Low-standard-standard GH: This group was randomized to receive 0.025 mg/kg/day of growth hormone for 7 doses given subcutaneously, followed by 2 weeks of wash out and then another 7 days of GH therapy (Nutropin AQ) at the standard dose of 0.05 mg/kg/day for 7 days.
- Standard- Low- Standard GH: This group was randomized to receive 0.05 mg/kg/day of growth hormone for 7 doses given subcutaneously followed by 2 weeks of wash out and then another 7 days of GH therapy (Nutropin AQ) at the low dose of 0.025 mg/kg/day for 7 days.
Period: First Intervention (7 Days)
Arm/Group | Low-standard-standard GH | Standard- Low- Standard GH
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Wash Out Period (2 Weeks)
Arm/Group | Low-standard-standard GH | Standard- Low- Standard GH
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Low-standard-standard GH | Standard- Low- Standard GH
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Standard Therapy of GH (12 Months)
Arm/Group | Low-standard-standard GH | Standard- Low- Standard GH
Started | 8 | 9
Completed | 6 | 8
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects will be randomized to either a low or standard arm. The low dose will get 0.025 mg/kg/day of growth hormone therapy and the standard dose arm will receive 0.05 mg/kg/dose given subcutaneously. After one week of therapy and 2 weeks of wash out, subjects will change the dose of GH therapy and will receive the alternate dose for another week. After that all subjects will be treated with the standard dose of GH therapy of 0.05 mg/kg/day for 6 months, re-evaluate growth velocity and then continue for another 6 months on GH.
Arm/Group | All Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.6 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: The Change in Amount of Insulin Like Growth Factor (IGF-I) Generated (Day 8-day 1)
Description: We will measure the amount of serum IGF-I generated after 7 days of growth hormone therapy (Day8-Day1).
Time Frame: Day 1 & Day 8
Measure: Mean (Standard Deviation); unit: mcg/L
Groups:
- Low Dose GH: Subjects will be randomized to either a low or standard arm. The low dose GH group will get 0.025 mg/kg/day of growth hormone therapy for 7 days followed by 2 weeks of wash out and then another 7 days of GH therapy on the standard dose of 0.05 mg/kg/dose given subcutaneously.
- Standard Dose GH: Subjects will be randomized to either a low or standard arm. The Standard dose GH group will get 0.05 mg/kg/day of growth hormone therapy for 7 days followed by 2 week wash out and then another 7 days of GH therapy on the low dose of 0.025 mg/kg/dose given subcutaneously.
Arm/Group | Low Dose GH | Standard Dose GH
Number analyzed (Participants) | 6 | 8
mcg/L | 115 (104) | 129 (112)

2. Secondary Outcome: Change in Height at 56 Weeks
Time Frame: week 1, week 56
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 14
cm | 10.3 (1.1)

ADVERSE EVENTS:
Groups:
- All Participants: There will be 2 arms in the study who will be randomized in a cross over design. The low dose will get 0.025 mg/kg/day of growth hormone therapy and the standard dose arm will receive 0.05 mg/kg/dose given subcutaneously. After one week of therapy and 2 weeks of wash out, subjects will change the dose of GH therapy and will receive the alternate dose for another week. After that all subjects will be treated with the standard dose of GH therapy of 0.05 mg/kg/day for 6 months.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Slow enrollment and the small number of participants in the study is the main limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less